CLINICAL TRIAL: NCT07269054
Title: Validation of the New Protocol Based on the Principles of the 1-repetition Maximum Test for Evaluating Maximum Respiratory Pressures in Individuals With Multiple Sclerosis.
Brief Title: Effects of Home-based Respiratory Muscle Training With New Load Adjustment Test in People With Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tamara del Corral Núñez-Flores (Other)
Collaborators: Ilustre Colegio Oficial de Fisioterapeutas de la Comunidad de Madrid (Unknown)
Responsible Party: Sponsor-Investigator, Tamara del Corral Núñez-Flores, Tenure-track professor with a PhD in the Department of Physiotherapy, Universidad Complutense de Madrid
Organization: Universidad Complutense de Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24/119-E_BC
Record Dates: First submitted 2025-11-19; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; Muscle Strength; Patient Outcome Assessment; Maximal Respiratory Pressures
MeSH Terms: conditions — Multiple Sclerosis | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory muscle training + 1-repetition maximum test (Experimental): Participants will perform an inspiratory and expiratory muscle training program by a threshold device at home, twice a day (morning inspiratory muscle training session and evening expiratory muscle training session) for 8 weeks supervised by a physiotherapist through a virtual platform. The load adjustment will be based on the principles of the 1-repetition maximum (RM) test.
  Interventions: Other: Respiratory muscle training + 1-repetition maximum test
- Respiratory muscle training + reference test (Active Comparator): Participants will perform an inspiratory and expiratory muscle training program by a threshold device at home, twice a day (morning inspiratory muscle training session and evening expiratory muscle training session) for 8 weeks supervised by a physiotherapist through a virtual platform. The load adjustment will be based on the conventional test to be performed during the 4th week.
  Interventions: Other: Respiratory muscle training + reference test

INTERVENTIONS:
Other: Respiratory muscle training + 1-repetition maximum test — Participants will engage in respiratory muscle training programme at home using a respiratory muscle training threshold device . This training will be conducted twice daily, five days a week, for eight weeks, with physiotherapist supervision provided by telerehabilitation. The load adjustment will be based on the principles of the 1-repetition maximum (RM) test.
  Arms: Respiratory muscle training + 1-repetition maximum test
Other: Respiratory muscle training + reference test — Participants will perform an inspiratory and expiratory muscle training program by a threshold device at home, twice a day (morning inspiratory muscle training session and evening expiratory muscle training session) for 8 weeks supervised by a physiotherapist through a virtual platform. The load adjustment will be based on the conventional test to be performed during the 4th week.
  Arms: Respiratory muscle training + reference test

SUMMARY:
The main objective of the present study is to verify whether respiratory muscle training programme (IMT+EMT; included both inspriratory and expiratory muscles with load adjustment based on the principles of the 1-repetition maximum (RM) test), applied by telerehabilitation, is an effective intervention (versus a respiratory muscle training programme (IMT+EMT; included both inspriratory and expiratory muscles with convetional load adjustment) in improving fragility, quality of life and physical function in people with Multiple Sclerosis.

DETAILED DESCRIPTION:
It is a single-blind randomized clinical trial study. Each participant will be randomly assigned to one of the following groups: 1) Inspiratory muscle training + Expiratory muscle training with load adjustment based on the principles of the 1-repetition maximum (RM) test , 2) Inspiratory muscle training + Expiratory muscle training with convetional load adjustment.

Each exercise training program will be applied twice (morning inspiratory muscle training session and evening expiratory muscle training session) per day 5 sessions per week during 8 weeks by a threshold device. The sessions will be supervised by a physiotherapist through a virtual platform.

Participants received baseline assessments at the beginning of the intervention, at the end of the 4th week (only the group 2), and post-intervention assessments at the end of the 8th week.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Multiple Sclerosis disease
* Age 18 years or older
* Clinical stability

Exclusion Criteria:

* Any condition that contraindicate respiratory muscle training
* Inability to close the lips to hold the training device's mouthpiece (e.g., facial paralysis)
* Pregnancy
* Inability to adhere to remote monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength | Pre -intervention and at the end of the respiratory muscle training (8 weeks)
  Maximal inspiratory preassure and Maximal expiratory preassure
Inspiratory muscle endurance | Pre -intervention and at the end of the respiratory muscle training (8 weeks)
  Inspiratory muscle endurance will be assed by an incremental load test that required subjects to breathe against inspiratory threshold loads that were increased each minute by 10% of baseline PI,max until voluntary task failure muscle endurance test. Inspiratory muscle endurance was defined as the PI,max sustained for a minimum of 1 min.

SECONDARY OUTCOMES:
Health related quality of life | Pre -intervention and at the end of the respiratory muscle training (8 weeks)
  To evaluate the health-related quality of life of the participants a valid, reliable and generic questionnaire will be used. EuroQol-five-dimensional Questionnaire a numerical value represented Health state as EQ-5D 'index values' or 'index scores' reflecting how good or bad a health state is. It consisted of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression), each of which has five severity levels that are described by statements appropriate to that dimension.
Fatigue | Pre -intervention and at the end of the respiratory muscle training (8 weeks)
  Modified Fatigue Impact Scale (MFIS). The MFIS is a valid and reliable instrument for assessing fatigue severity. It consists in 21 items. Higher scores mean a worse fatigue.
Fragility | Pre -intervention and at the end of the respiratory muscle training (8 weeks)
  Frailty indexes (FI) and the Comprehensive GeriatricAssessment (CGA) are multidimensional tools. FI serve to quantitatively measure frailty levels. They have shown to have an excellent correlation with mortality.
Degree of disability | Pre -intervention and at the end of the respiratory muscle training (8 weeks)
  The Barthel index (BI) is a 10-item activities of daily living ordinal scale used primarily for disability measurement. The values assigned to each item are based on the time and amount of physical assistance required for a patient to perform a common daily activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Asociación Mostoleña de Esclerosis Múltiple, Móstoles, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No